CLINICAL TRIAL: NCT03940716
Title: M-Health to Decrease Youth Substance Misuse & High-Risky Illegal Firearm Behaviors
Brief Title: Project IntERact Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Patrick Carter, Assistant Professor of Emergency Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00104549; K23DA039341 (NIH)
Record Dates: First submitted 2019-04-30; First posted 2019-05-07 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Violence; Substance Use; Criminal Behavior
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IntERact (Experimental): Participants randomized to this condition will receive behavioral therapy comprised of motivational interviewing, cognitive behavioral skills therapy, and care management. Youth will receive a total of six sessions, one delivered in the emergency department at the time of recruitment and five delivered over the five subsequent weeks after the ED visit (i.e., baseline). Participants will also receive a smartphone APP that will deliver intervention content between therapy sessions, including tailored MI+CBT messages (tailored by daily survey responses), one-touch pro-social contact, psycho-educational materials, GPS-enabled "just-in-time" tailored alerts, and facilitated access to care management resources.
  Interventions: Behavioral: IntERact
- Enhanced Usual Care Condition (No Intervention): Participants randomized to this condition will receive a pamphlet with violence, mental health, and substance use resources.

INTERVENTIONS:
Behavioral: IntERact — This intervention integrates motivational interviewing, cognitive behavioral skills therapy, and care management into a single behavioral counseling intervention delivered by a therapist. The intervention is delivered either in the emergency department or remotely over the subsequent 5 weeks for a total of six therapy sessions (~30 min each). A smartphone app is also loaded on the participant's phone and delivers additional behavioral intervention content, including tailored MI+CBT messages (tailored by daily survey responses), one-touch pro-social contact encouragement, psycho-educational materials, GPS-enabled "just-in-time" tailored alerts, and facilitated access to care management resources.
  Arms: IntERact

SUMMARY:
This study will use a randomized control trial design (RCT) to pilot test a multisession remote therapy behavioral intervention for risky firearm behaviors and associated behaviors/consequences among adolescents. The study will pilot a state-of-the-art intervention delivery approaches (e.g., remote therapy, smartphone-based APP intervention content delivery) for reducing violence and associated behaviors among urban youth. Given the significant morality and mortality associated with firearm violence, the study will have significant impact by identifying optimal intervention strategies for future large-scale behavioral intervention trials.

DETAILED DESCRIPTION:
The specific aim of this pilot study is to pilot test an m-health intervention, as compared to enhanced usual care [n=70; 35/group], with eligible youth to assess intervention acceptability, feasibility, and fidelity, as well as trends towards decreased risky firearm behaviors, substance use, and criminal justice involvement. Specifically, 70 youth (ages 16-24) in the ED screening positive for firearm carriage and smartphone ownership will be randomly assigned (stratified by age/gender) to either the IntERact group or the control group. IntERact group participants will receive an Emergency Department (ED) session of behavioral therapy, followed by five additional remote therapy sessions of behavioral therapy delivered over the 5 weeks following their ED visit. Behavioral therapy will be comprised of motivational interviewing (MI), cognitive behavioral therapy (CBT), and strengths-based care management (CM). In addition, youth in the IntERact group will also receive a smartphone APP that will be downloaded to their phone. The APP will deliver daily surveys, daily tailored MI and CBT messages in response to survey results, one-touch access to pro-social supports, psycho-educational materials, GPS-enabled message alerts, and facilitated access to CM resources. Youth enrolled in the control group will receive a pamphlet with local violence, substance use, and mental health resources. A follow-up assessment will be completed in each group at 4 months post-ED visit. Pilot data will aid in refining and clarifying content and clinical trial design elements for a future fully powered randomized control trial of the intervention (i.e., R01 proposal).

ELIGIBILITY:
Inclusion Criteria:

* Past 4-month firearm carriage
* Ownership of a smartphone with APP capabilities

Exclusion Criteria:

* Non-english speaking patients
* Patients unable to provide informed consent due to mental incompetence, incarceration (i.e., active police custody), medically unstable (abnormal vital signs requiring urgent resuscitation)
* Patients presenting for acute suicidal ideation or acute suicide attempt, child abuse or sexual assault.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Acceptability: enrollment rates | Baseline
  Acceptability will be measured at baseline using study enrollment rates
Participant Satisfaction (Helpfulness/Likability) | Baseline to 4-month follow-up
  Participant satisfaction measures of helpfulness and likability will be assessed for individual intervention sessions and content (measured during post-tests after each session and at the 4-month follow-up).
  Measures have been used in prior work (Walton 2010) and each item is scored on a 5-point likert scale (1=not at all; 5=extremely) with % of enrolled patients who completed sessions reporting scores of 4 or 5 reporting high likability or helpfulness.
Feasibility of Daily Assessments: completion rates of daily assessments | Baseline to Post-Intervention (~5 weeks)
  Feasibility will be measured during the course of the study by examining completion rates of daily assessments.
Feasibility of Remote Sessions: Completion rates for Remote Therapy Sessions | Baseline to Post-Intervention (~5 weeks)
  Completion rates for Remote Therapy Sessions
Feasibility of 4-month follow-ups: % of eligible enrolled youth who complete follow-up | 4-month Follow-up
  Completion rates for 4-month follow-up assessments (i.e., % of eligible enrolled youth who complete follow-up).
Fidelity | Baseline to 4-month Follow-up
  Fidelity will be measured using standard therapy adherence measures coding audio tapings of remote therapy sessions.

SECONDARY OUTCOMES:
Change in Risky Firearm Behaviors | Baseline to 4-month Follow-up
  Composite measure used in prior work (Carter 2019). Composite measure uses items from the Tulane University Youth Study and Conflict Tactics Scale capturing frequency and severity of firearm-related behaviors (e.g., carriage, threats, use, etc.). Items will be summed to create a summary score.

CONTACTS AND LOCATIONS:
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT03940716/ICF_000.pdf